CLINICAL TRIAL: NCT07285681
Title: Effectiveness of Neurofeedback in Treatment of Attention Deficit Hyperactivity Disorder in a Sample of Patients in Tanta, Egypt
Brief Title: Neurofeedback in Treatment of Attention Deficit Hyperactivity Disorder
Acronym: ADHD NF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Ahmed Salem, Lecturer of Neuropsychiatry - Faculty of Medicine - Tanta University, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR1295/7/25
Record Dates: First submitted 2025-10-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: All participants in this study will be subjected to the following
  1. Collection of socio demographic data using El Gilany and El Wasify scale
  2. The Conners Rating Scale For ADHD
     * Performed at base line before starting neurofeedback
     * After 15 sessions follow up
     * After ending the sessions
  3. Neurofeedback:
     * The patients will receive 30 sessions each lasting 50 minutes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effectiveness of Neurofeedback in treatment of Attention Deficit Hyperactivity Disorder (Experimental): 3- Neurofeedback:
  - The patients will receive 30 sessions each lasting 50 minutes.
  Interventions: Device: Neurofeedback

INTERVENTIONS:
Device: Neurofeedback — The aim of this study to assess the effectiveness of Neurofeedback in management of Attention Deficit Hyperactivity Disorder in a sample of patients in Tanta city, Egypt

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a common , chronic , and debilitating disorder . Although pharmacological treatments for ADHD can be easily implemented and are usually effective, their long-term therapeutic effects are still uncertain and adverse events are common, especially sleep problems, decreased appetite, and growth deceleration. Furthermore, psychosocial treatments, such eas parental training and behavioral therapy seem to be effective only during its delivery, and their effects are rarely sustained long-term .

Neurofeedback is a biofeedback method based on the rationale that there is a relationship between surface EEG and the underlying thalamocortical mechanisms responsible for its rhythms and frequency modulations .

Variations in alertness and behavioural control appear directly related to thalamocortical generator mechanisms. The principle of NF is that over time, participants learn operant control of their EEG and change from an "abnormal" state to one resembling that of typically developing children. This process is thought to eventually remediate the symptoms associated with ADHD .

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a common , chronic , and debilitating disorder . Although pharmacological treatments for ADHD can be easily implemented and are usually effective, their long-term therapeutic effects are still uncertain and adverse events are common, especially sleep problems, decreased appetite, and growth deceleration. Furthermore, psychosocial treatments, such eas parental training and behavioral therapy seem to be effective only during its delivery, and their effects are rarely sustained long-term Clinical guidelines for attention-deficit/hyperactivity disorder (ADHD) recommend multimodal treatment approaches, with current evidence suggesting that medication, including methylphenidate and various amphetamine formulations, in conjunction with psychosocial treatment are most effective in the short-term . Medication treatments have large effect size in the acute treatment of ADHD and, when combined with psychosocial treatments, large effects up to 2 years of treatment were observed. Nevertheless, it is widely accepted that further treatments with long-lasting effects have to be developed and evaluated .

Over the last decade, an increasing number of studies investigating non-pharmacological treatments have been published. Neurofeedback (NF), which aims at improving self-regulation of brain activity (most often the electroencephalogram, EEG) using a brain-computer interface, has gained popularity. A promising aspect of neurofeedback is that it may rely on procedural learning, thereby potentially allowing lasting effects and thus longer clinical benefit after completion of neurofeedback treatment In recent years, several randomized control studies (RCTs) and meta-analyses have been published on the efficacy of neurofeedback for children with ADHD, overall with mixed results and interpretations .

Neurofeedback is a biofeedback method based on the rationale that there is a relationship between surface EEG and the underlying thalamocortical mechanisms responsible for its rhythms and frequency modulations .

Variations in alertness and behavioural control appear directly related to thalamocortical generator mechanisms. The principle of NF is that over time, participants learn operant control of their EEG and change from an "abnormal" state to one resembling that of typically developing children. This process is thought to eventually remediate the symptoms associated with ADHD The aim of this study to assess the effectiveness of Neurofeedback in management of Attention Deficit Hyperactivity Disorder in a sample of patients in Tanta city, Egypt

All participants in this study will be subjected to the following

1. Collection of socio demographic data using El Gilany and El Wasify scale
2. The Conners Rating Scale For ADHD

   * Performed at base line before starting neurofeedback
   * After 15 sessions follow up
   * After ending the sessions
3. Neurofeedback:

   * The patients will receive 30 sessions each lasting 50 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between 12- 18 years old
* Both sexes are included (males & females).
* Willingness to participate to complete study procedures

Exclusion Criteria:

* Unwilling to participate in the study.
* Other Psychiatric disorders.
* Intellectual disability

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
5. The Arabic version of Conners Rating Scale | At the baseline after 35 days after 70 days
  The Arabic version of Conners' Rating Scale was developed as a comprehensive checklist for acquiring parental reports of the basic presenting problems for children referred to an outpatient psychiatric setting .The Conners' Comprehensive Behavior Rating Scale is a questionnaire that focuses on behavioral, social, and academic issues in children and adolescents. It can help diagnose & rate attention deficit hyperactivity disorder .The Arabic version of Conners' Rating scale is composed of 48 items divided on 6 scales. The 6 scales include: conduct disorder, learning problems, psychosomatic problems, impulsivity, hyperactivity & anxiety
  It is usually considered normal when scores are less than 60, while scores above 60 are signs of academic, behavioral, or social issues. There are several different classes as well:
  * A T -score of more than 60 can indicate that the child may have an issue such as ADHD.
  * A T-score greater than 60 but under 70 may indicate moderately severe issues.
Collection of socio demographic data using El gilany and ElWasify scale | - Performed at base line
  Socioeconomic status(SES) is measured by 3 variables: education, occupation and income. While SES has been seen as an inherited factor, in modern society it may migrate on the basis of factors such as occupation, education, income, type of housing, material possessions. The final scale included 7 domains in the form of education , occupation, family, family possession, home sanitation, health care and economic domain with a total score of 84, with a higher score indicating better SES,

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroPsychiatry Department - Faculty of Medicine - Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No